CLINICAL TRIAL: NCT01587365
Title: Randomized, Double-Blind, Placebo-Controlled, Ascending Single-Dose Study to Evaluate the Safety, Pharmacokinetics and Pharmacodynamics of BMS-962476 in Healthy Subjects and in Patients With Hypercholesterolemia on Statin Therapy
Brief Title: Single Ascending Dose Safety Study of BMS-962476 in Healthy Subjects and Patients With Elevated Cholesterol on Statins
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: CV206-001
Record Dates: First submitted 2012-04-26; First posted 2012-04-30 (Estimated); Last update posted 2013-09-04 (Estimated); Status verified 2013-09

CONDITIONS: Atherosclerosis
MeSH Terms: conditions — Atherosclerosis | interventions — BMS-962476

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (8):
- Panel 1: BMS-962476 SC (0.01 mg/Kg) or Placebo (Experimental): BMS-962476 0.01 mg/kg or Placebo matching with BMS-962476 0 mg liquid subcutaneously (SC), Single Dose, 1 day
  Interventions: Biological: BMS-962476; Biological: Placebo matching with BMS-962476
- Panel 2: BMS-962476 SC (0.03 mg/Kg) or Placebo (Experimental): BMS-962476 0.03 mg/kg or Placebo matching with BMS-962476 0 mg liquid subcutaneously (SC), Single Dose, 1 day
  Interventions: Biological: BMS-962476; Biological: Placebo matching with BMS-962476
- Panel 3: BMS-962476 SC (0.1 mg/Kg) or Placebo (Experimental): BMS-962476 0.1 mg/kg or Placebo matching with BMS-962476 0 mg liquid subcutaneously (SC), Single Dose, 1 day
  Interventions: Biological: BMS-962476; Biological: Placebo matching with BMS-962476
- Panel 4: BMS-962476 SC (0.3 mg/Kg) or Placebo (Experimental): BMS-962476 0.3 mg/kg or Placebo matching with BMS-962476 0 mg liquid subcutaneously (SC), Single Dose, 1 day
  Interventions: Biological: BMS-962476; Biological: Placebo matching with BMS-962476
- Panel 5: BMS-962476 IV (0.3 mg/Kg) or Placebo (Experimental): BMS-962476 0.3 mg/kg or Placebo matching with BMS-962476 0 mg liquid intravenously (IV), Single Dose, 1 day
  Interventions: Biological: BMS-962476; Biological: Placebo matching with BMS-962476
- Panel 6: BMS-962476 IV (1.0 mg/Kg) or Placebo (Experimental): BMS-962476 1.0 mg/kg or Placebo matching with BMS-962476 0 mg liquid intravenously (IV), Single Dose, 1 day
  Interventions: Biological: BMS-962476; Biological: Placebo matching with BMS-962476
- Panel 7: Statin + BMS-962476 SC (0.1 mg/Kg) or Placebo (Experimental): BMS-962476 0.1 mg/kg or Placebo matching with BMS-962476 0 mg liquid subcutaneously (SC), Single Dose, 1 day
  Interventions: Biological: BMS-962476; Biological: Placebo matching with BMS-962476
- Panel 8: Statin + BMS-962476 SC (0.3 mg/Kg) or Placebo (Experimental): BMS-962476 0.3 mg/kg or Placebo matching with BMS-962476 0 mg liquid subcutaneously (SC), Single Dose, 1 day
  Interventions: Biological: BMS-962476; Biological: Placebo matching with BMS-962476

INTERVENTIONS:
Biological: BMS-962476
Biological: Placebo matching with BMS-962476

SUMMARY:
To obtain safety and tolerability information in healthy subjects is administered as a single dose

DETAILED DESCRIPTION:
* Study Classification: Pharmacokinetics and Pharmacodynamics
* Intervention Model: Single Ascending Dose (SAD) study
* Allocation: Randomized Non-Stratified

ELIGIBILITY:
Inclusion Criteria:

* Healthy population

  * Untreated low density lipoprotein cholesterol (LDL-c) ≥ 130 and ≤ 190 mg/dL and triglycerides ≤ 200 mg/dL
  * Body Mass Index (BMI) of 18 to 35 kg/m2 inclusive
  * Men and women, ages 18 to 65 years, inclusive
* Statin population

  * Patients with hypercholesterolemia on stable statin therapy for 6 weeks prior to enrollment
  * At enrollment, LDL-c ≥ 100mg/dL and triglycerides ≤ 200 mg/dL
  * Patients with controlled hypertension on a stable dose of no more than two antihypertensive drugs
  * BMI of 18 to 37 kg/m2 inclusive
  * Men and women, ages 18 to 75 years inclusive

Exclusion Criteria:

* Healthy Population

  * Subjects with fasting LDL-c < 130 or > 190 mg/dL, or fasting triglycerides > 200 mg/dL
  * Subjects at increased 10-year cardiovascular risk of ≥ 20% based on Framingham risk score
  * Subjects with any significant acute or chronic medical illness at the time of screening, including history of cancer, known history of sickle cell disease or trait, and known history of thalassemia
* Statin population

  * Patients with fasting LDL-c < 100mg/dL, or fasting triglycerides > 200 mg/dL on statin therapy
  * Patients on prescription or over the counter lipid-lowering therapy other than statin therapy
  * Patients with established atherosclerotic vascular disease
  * Patients with diabetes who are requiring oral or injectable anti-diabetic drug therapy
  * Patients with uncontrolled hypertension or controlled hypertension requiring more than two antihypertensive drugs
  * Patients with any significant acute or chronic medical illness that is severe, progressive or uncontrolled at the time of screening
* Use of any lipid lowering medication including over the counter products (eg, niacin > 500 mg; omega-3 fatty acids > 1000 mg; red rice yeast; phytosterols or stanol esters) for lipid lowering within 30 days prior to screening visit (42 days for fibrates) with the exception of stable statin therapy in the target disease population
* Prior treatment with any monoclonal antibody or investigational protein biologic within the preceding one year before study drug administration
* Concurrent or use within 3 months of study drug administration of marketed or investigational systemic or inhaled corticosteroids or other immunosuppressant drugs, and within 6 weeks for topical corticosteroids

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2012-05; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of BMS-962476 as measured by the number of subjects with serious adverse events, deaths or discontinuations due to adverse events (AEs), AEs of injection site reactions, or potentially clinically significant changes in vital signs | Up to Day 43

SECONDARY OUTCOMES:
Pharmacodynamic effects of single subcutaneous (SC) and intravenous (IV) doses of BMS-962476 | Up to Day 43
  Pharmacodynamic effects will be measured by fasting lipid panel
Maximum observed plasma concentration (Cmax) of single dose pharmacokinetics (PK) and dose proportionality of BMS-962476 following SC and IV administration | 17 time points up to Day 43
Time of maximum observed plasma concentration (Tmax) of single dose pharmacokinetics (PK) and dose proportionality of BMS-962476 following SC and IV administration | 17 time points up to Day 43
Area under the plasma concentration-time curve from time zero to the time of last quantifiable plasma concentration [AUC(0-T)] of single dose pharmacokinetics (PK) and dose proportionality of BMS-962476 following SC and IV administration | 17 time points up to Day 43
Area under the plasma concentration-time curve from time zero extrapolated to infinite time [AUC(INF)] of single dose pharmacokinetics (PK) and dose proportionality of BMS-962476 following SC and IV administration | 17 time points up to Day 43
Plasma elimination half-life (T-HALF) of single dose pharmacokinetics (PK) and dose proportionality of BMS-962476 following SC and IV administration | 17 time points up to Day 43
Total body clearance (CL/F) of BMS-962476 SC Dosing | 15 time points up to Day 43
Total body clearance (CL) of BMS-962476 IV Dosing | 17 time points up to Day 43
Volume of distribution at steady state (Vss/F) of BMS-962476 SC Dosing | 15 time points up to Day 43
Volume of distribution at steady state (Vss) of BMS-962476 IV Dosing | 15 time points up to Day 43
Absolute bioavailability (F) of total and free BMS-962476 | 15 time points up to Day 43
Frequency of anti-BMS-962476 antibodies (immunogenicity) following single SC and IV doses of BMS-962476 | Up to Day 43

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Metabolic And Atherosclerosis Research Center/ Medpace Clinical Pharmacology, Cincinnati, Ohio, United States

REFERENCES:
- See also: BMS clinical trial educational resource — http://www.bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx